CLINICAL TRIAL: NCT01193543
Title: Effect of Calanus Oli on Intra-abdominal Fat, Glucose Tolerance and Lipids in Man
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UIT-ENDO-2010-4
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- calanus oil (Experimental): calanus oil 1 gram twice daily
  Interventions: Dietary Supplement: calanus oil
- olive oil (Placebo Comparator): olive oil 1 gram twice daily
  Interventions: Dietary Supplement: olive oil

INTERVENTIONS:
Dietary Supplement: calanus oil — 1 gram twice daily
  Arms: calanus oil
Dietary Supplement: olive oil — 1 gram twice daily
  Arms: olive oil

SUMMARY:
Preliminary studies in rats and mice indicate that calanus oil reduce accumulation of intra-abdominal fat. Pilot studies in humans have shown no adverse effects. In the present study 120 subjects, males and females, 20-65 years old, BMI 25-30 kg/m2 will be included and given calanus oli 1 g twice daily versus placebo for 1 year. The hypothesis is that calanus oil will reduce intra-abdominal fat, improve glucose tolerance and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 25-30 kg/m2
* age 20-65 years

Exclusion Criteria:

* diabetes
* coronary heart disease last 12 months
* unstable angina pectoris
* cancer diagnosed the last 5 years
* use of lipid lowering drugs
* seafood allergy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Intra-abdominal fat as measured with CT scan | at the end of 12 months intervention

SECONDARY OUTCOMES:
oral glucose tolerance test | at the end of 12 months intervention
lipid status | at the end of 12 months intervention
systolic and diastolic blood pressure | at the end of 12 months intervention
markers of inflammation - C-reactive protein (CRP) | at the end of 12 months intervention
body weight | at the end of 12 months intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Jorde, Professor, Principal Investigator — University of Tromso
Locations (1):
- University of Tromso, Tromsø, Norway